CLINICAL TRIAL: NCT02591355
Title: A Monocentric, Double-blind, Randomized, Active- and Placebo-controlled Split-scalp Study to Evaluate the Clinical Effectiveness of Platelet-rich Plasma (PRP) in the Treatment of Androgenetic Alopecia
Brief Title: Evaluate the Clinical Effectiveness of RegenKit Platelet-rich Plasma (PRP) in Androgenetic Alopecia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regen Lab SA (Industry)
Collaborators: RegenLab USA LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RL 03
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Androgenetic Alopecia
Keywords: Platelet Rich Plasma; Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Autologous Platelet Rich Plasma (Experimental): Autologous Platelet Rich Plasma injection
  Interventions: Device: Autologous Platelet Rich Plasma
- Saline (Placebo Comparator): Saline solution injection
  Interventions: Device: Saline solution injection

INTERVENTIONS:
Device: Autologous Platelet Rich Plasma — Autologous Platelet Rich Plasma a novel therapeutic modality used in numerous applications. In dermatology, its uses have included treatment of chronic wounds and facial rejuvenation. More recently, anecdotal reports have suggested some efficacy in the treatment of hair loss.
  Arms: Autologous Platelet Rich Plasma
Device: Saline solution injection — Placebo is a saline solution
  Arms: Saline

SUMMARY:
Platelet rich plasma (PRP) therapy is a novel therapeutic modality that has seen broad applications for a number of medical indications including those in orthopedics, dentistry, and dermatology. In dermatology, its uses have included treatment of chronic wounds and facial rejuvenation. More recently, anecdotal reports have suggested some efficacy in the treatment of hair loss, but to the best of our knowledge, there has been only one published case series documenting its use for this indication.

DETAILED DESCRIPTION:
This study was designed to better assess the efficacy of PRP in hair loss, we therefore propose to study interval intralesional PRP injections for patients with androgenetic alopecia (AGA). Androgenetic alopecia is the most common form of hair loss world-wide. Although there are currently numerous treatment options for this indication including minoxidil, 5-alpha reductase inhibitors and follicular unit transplant, many of the medical treatment options have undesirable side effects, particularly in women of child bearing age. These well-documented adverse reactions include impotency, hypertrichosis, and birth defects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18-60 with AGA
* Completed informed consent form
* Ludwig stage 1-2 for women
* Norwood Hamilton Stage 3 to 5 for men

Exclusion Criteria:

* Pregnancy or breastfeeding
* Younger than 18 years
* Uses of minoxidil and/or 5-alpha reductase inhibitors (such as finasteride or dutasteride) within 3 months of enrolling in the study
* History of hair transplantation
* Use of any cosmetic product aimed at improving or correcting the signs of hair loss within 2 weeks prior to screening
* Facial cancer (squamous and basal cell carcinoma, melanoma)
* Hereditary or acquired hematologic/coagulation disorders such as: platelet dysfunction syndrome, critical thrombocytopenia, hypofibrinogenemia, impaired coagulation, drepanocytosis (sickle cell anemia).
* Hemodynamic instability
* Acute infection
* Auto-immune disease such as Hashimoto, rheumatoid arthritis, or lupus (exception: vitiligo and alopecia areata)
* Malignancy with or without metastatic disease
* Chemotherapy
* Dermatological diseases affecting the face (e.g. porphyria)
* Anticoagulant therapy
* Patients taking Aspirin or other NSAIDs (Nonsteroidal anti-inflammatory drugs) such as Nurofen, Voltaren, Diclofenac or Naproxen can participate, provided medication is interrupted 7 days before beginning of the treatment
* Patients taking vitamin E supplements can participate, provided medication is interrupted 14 days before beginning of the treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the changes in hair density of androgenetic alopecia | 5 months
  Evaluate split scalp changes in hair density of androgenetic alopecia after 5 month treatment of Autologous Platelet Rich Plasma prepared with the RegenBCT-1 kit compared to other half of the scalp treated with saline solution.

SECONDARY OUTCOMES:
Evaluate the changes of hair diameter and hair shedding in androgenetic alopecia | 5 months
  Evaluate the changes of hair diameter and hair shedding in androgenetic alopecia after 5 months treatment of Autologous Platelet Rich Plasma prepared with the RegenBCT-1 kit compared to other half of the scalp treated with saline solution.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Shapiro, MD, Principal Investigator — NYU School of Medicine, Langone Medical Center, New-York University
Locations (2):
- United States (2):
  - Axis Clinical Trials, Los Angeles, California
  - NYU Dermatologic Associates, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided